CLINICAL TRIAL: NCT01525732
Title: Prospective Study on the Feasibility and Effectiveness of Per-Oral Endoscopic Myotomy (P.O.E.M.) for Treatment of Primary Esophageal Motility Disorders
Brief Title: Per-Oral Endoscopic Myotomy (P.O.E.M.) for Treatment of Esophageal Motility Disorders
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan Chiu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2010_430
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Achalasia; Hypertensive LES
Keywords: Achalasia, Hypertensive LES
MeSH Terms: conditions — Esophageal Achalasia

ARMS (1):
- POEM (Other): Per Oral Endoscopic Myotomy
  Interventions: Procedure: Per Oral Endoscopic Myotomy

INTERVENTIONS:
Procedure: Per Oral Endoscopic Myotomy

SUMMARY:
Spastic esophageal motility disorders induced significant symptoms including dysphagia, retrosternal pain and regurgitation. Per oral endoscopic myotomy (P.O.E.M.) is a novel approach to perform myotomy through the esophagus with long submucosal tunnel. This study aimed to investigate the feasibility and safety of P.O.E.M. and translate the techniques from animal study to clinical practice in human.

ELIGIBILITY:
Inclusion Criteria:

* All patients with age ranged 18 to 80 who had primary esophageal motility disorders will be recruited. The primary motility disorders included: Achalasia, hypertensive LES, Nutcracker esophagus and Diffuse esophageal spasm.

Exclusion Criteria:

* Patients will be excluded from this study with the followings -

  1. Pregnancy
  2. Informed consent not available
  3. Previous history of esophagectomy or mediastinal surgery
  4. Previous history of endoscopic resection for early esophageal cancers, including endoscopic mucosal resection and endoscopic submucosal dissection
  5. End-stage Achalasia with dilated esophagus more than 6cm on Barium swallow

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Dysphagia score before and after P.O.E.M. | From 1st day after POEM to within 2 weeks after POEM

SECONDARY OUTCOMES:
Eckardt score before and after P.O.E.M. | Before and 1 month after POEM
Post-operative pain | From Day 1 to until 2 weeks after POEM
Operative time | Up to 24 hours
Hospital stay | From day of admission till up to 30 days
Perioperative complication | 30 days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chiu PW, Wu JC, Teoh AY, Chan Y, Wong SK, Liu SY, Yung MY, Lam CC, Sung JJ, Chan FK, Lau JY, Ng EK. Peroral endoscopic myotomy for treatment of achalasia: from bench to bedside (with video). Gastrointest Endosc. 2013 Jan;77(1):29-38. doi: 10.1016/j.gie.2012.08.018. Epub 2012 Oct 6. PMID 23043852